CLINICAL TRIAL: NCT06219473
Title: Efficacy of Fascia Lata Allograft and Platelet Rich Fibrin Versus Connective Tissue Graft on the Periodontal Phenotype Around Dental Implant in Upper Anterior Region: A Randomized Controlled Clinical Trial
Brief Title: Efficacy of Fascia Lata Allograft and Platelet Rich Fibrin on the Periodontal Phenotype Around Dental Implant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Radwan Elhadidy, assistant lecturer at Delta university for science and technology, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-87
Record Dates: First submitted 2024-01-03; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Allograft
Keywords: Fascia lata allograft

STUDY DESIGN:
Intervention Model Description: Patients were classified into three main groups:
  Group 1 (Study group) It includes eight patients seeking for implant placement in the upper anterior areas and implants will be placed with the application of fascia lata allograft membrane.
  Group 2 (Study group) It includes eight patients seeking for implant placement in the upper anterior area and implants will be placed with the application of PRF.
  Group 3 (Control group) It includes eight patients seeking for single implant placement at the upper anterior area and those patients will be received their implants with subepithelial connective tissue graft.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fascia Lata (Study group) (Experimental): It includes eight patients seeking for implant placement in the upper anterior areas and implants will be placed with the application of fascia lata allograft membrane.
  Interventions: Drug: Fascia lata membrane
- PRF (Study group) (Experimental): It includes eight patients seeking for implant placement in the upper anterior area and implants will be placed with the application of PRF.
  Interventions: Drug: Platlet Rich fibrin membrane
- Connective tissue Graft(Control group) (Active Comparator): It includes eight patients seeking for single implant placement at the upper anterior area and those patients will be received their implants with subepithelial connective tissue graft.
  Interventions: Drug: subepithelial connective tissue graft

INTERVENTIONS:
Drug: Fascia lata membrane — novel allogenic derived acellular matrix produced from human fascia lata allograft
  Other Names: Fascia lata allograft
  Arms: Fascia Lata (Study group)
Drug: Platlet Rich fibrin membrane — Platelet-rich fibrin (PRF) or leukocyte- and platelet-rich fibrin (L-PRF) is a derivative of PRF where autologous platelets and leukocytes are present in a complex fibrin matrix to accelerate the healing of soft and hard tissue
  Other Names: Platlet Rich fibrin
  Arms: PRF (Study group)
Drug: subepithelial connective tissue graft — The connective tissue is generally taken from the hard palate, although it may be taken from other sites as well, such as the maxillary tuberosity area.
  Other Names: Connective tissue graft
  Arms: Connective tissue Graft(Control group)

SUMMARY:
To compare between the efficacy of fascia lata allograft and platelet rich fibrin versus subepithelial connective tissue graft on periodontal phenotype (thickness and width of keratinized tissue, labial bone thickness) around dental implant in upper anterior region.

DETAILED DESCRIPTION:
In order to evaluate the effectiveness of fascia lata allograft, platelet-rich fibrin, and subepithelial connective tissue graft on periodontal phenotype (including the thickness and width of keratinized tissue, as well as the thickness of labial bone) around dental implants in the upper anterior region, the purpose of this study is to compare the three types of grafts.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with thin gingival biotype (gingival thickness was ≤1 mm)
2. The height of keratinized gingiva for the site selected should be ≥2 mm.
3. Ability to maintain good oral hygiene as evidenced in recall visits.

Exclusion Criteria:

1. Smoker patient and pregnant or lactating woman.
2. Patient with poor oral hygiene or active periodontal disease.
3. Traumatic occlusion or para-functional habits such as clenching or bruxism.
4. Patient with limited mouth opening

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients age ranged from 20 to 50
Enrollment: 24 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Pink aesthetic score | 6 Months
  Pink esthetic score The gingival response to a anterior esthetic evaluation is assessed by the Pink Esthetic Score (PES) from clinical photography

CONTACTS AND LOCATIONS:
Overall Officials: Enas elgendy, Prof, Study Chair — Professor of Oral medicine and Periodontology at Kafr Elsheikh University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moraschini V, Kischinhevsky ICC, Sartoretto SC, Shibli JA, Dias AT, Sacco R, Yates J, Calasans-Maia MD. Is there any biomaterial substitute for peri-implant soft tissue phenotype modification? A network meta-analysis of the appraisal literature. Int J Oral Maxillofac Surg. 2022 Apr;51(4):526-534. doi: 10.1016/j.ijom.2021.07.005. Epub 2021 Aug 7. PMID 34373184

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT06219473/Prot_SAP_000.pdf